CLINICAL TRIAL: NCT06147011
Title: Development of 3D Printing High-Fidelity Thyroid Fine Needle Aspiration Exam Medical Education Model to Facilitate Student Learning and Practice
Brief Title: 3D Thyroid Education Model for Student
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FJUH111215-2
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Satisfaction, Personal
Keywords: 3D printing; medical education model; high-fidelity simulation; thyroid; fine needle aspiration
MeSH Terms: conditions — Personal Satisfaction; Thyroid Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D medical education model group (Experimental): Received a regular learning plus 3D printing model
  Interventions: Other: 3D printed educational model

INTERVENTIONS:
Other: 3D printed educational model — Slide-based presention plus 3D printed thyroid fine needle aspiration model

SUMMARY:
The purpose of our study is to develop a high-fidelity thyroid education model, that can be utilized for medical students/ PGY doctors/ residents training. This model can help them better understand the structure of thyroid, learn about what are thyroid nodules, and practice thyroid fine needle aspiration examination with the model. The investigators would also evaluate the efficacy of using this model in student teaching.

DETAILED DESCRIPTION:
Background： Thyroid nodular disorder is prevalent in Endocrine clinics, and while thyroid fine needle aspiration examination is crucial for evaluating nodules, conveying the procedure to students is challenging. The investigators propose a high-fidelity 3D model to enhance education, especially for hands-on practice. Our study aims to assess the model's education efficacy.

Study Design： This is a prospective study.

Methods： In our study, 3D scanning and 3D printing technology will be used to create the thyroid high-fidelity model. The investigators plan to choose 3D printing materials that enable the practice of thyroid fine needle aspiration produce with No.22 or No.23 needles.

Effect： The investigators hope to assist students understand the structure of thyroid and thyroid nodules better. And students will be able to practice thyroid fine needle aspiration examination with the 3D high-fidelity model. The outcome of our study may be utilized in medical schools or hospitals to facilitate student education.

Key words： 3D printing; medical education model; high-fidelity simulation; thyroid; fine needle aspiration

ELIGIBILITY:
Inclusion Criteria:

* Medical students, medical interns, PGY physicians, and resident physicians training at Fu Jen Catholic University Hospital

Exclusion Criteria:

* Refused to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient education effectiveness questionnaire | immediately after the intervention
  higher means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No